CLINICAL TRIAL: NCT07237776
Title: Effect of Virtual Reality in Abdominal Muscle Recovery After Cesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Heba Alaa Eid Abd-Elhafez, Lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/2111/MTI.PT/2409241
Record Dates: First submitted 2025-08-28; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Cesarean Section Complications

STUDY DESIGN:
Intervention Model Description: Randomized control trial
Who Masked: Participant
Masking Description: single blind participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- virtual reality group (Experimental): using virtual reality technology to perform abdominal muscle training 3 sessions per week for eight weeks
  Interventions: Device: Virtual reality Glasses
- Active Abdominal exercise group (Experimental): abdominal muscle training using Active Abdominal exercises 3 sessions per week for eight weeks.
  Interventions: Other: active abdominal exercises

INTERVENTIONS:
Device: Virtual reality Glasses — Virtual reality Glasses (is an advanced, standalone virtual reality (VR) headset that delivers a fully immersive experience without reliance on external hardware such as a PC, gaming console, or external tracking sensors. It utilizes an integrated inside-out tracking system that enables users to move freely within their physical environment while maintaining accurate spatial orientation. The device incorporates high-resolution displays, a high-performance processor, and ergonomically designed controllers that enhance interactivity and user engagement within virtual environments
  Arms: virtual reality group
Other: active abdominal exercises — Trunk flexion refers to bending the spine forward, mainly activating the rectus abdominis (the "six-pack" muscle). This movement is commonly seen in crunches or sit-ups.
  Straight Leg Raise (SLR) is a movement that strengthens the lower abdominal muscles and hip flexors. It involves raising the legs while keeping them straight, without bending at the knees. both exercises were done with 30 reptations (3 sessions per week for 8 weeks)
  Arms: Active Abdominal exercise group

SUMMARY:
Cesarean section is mainly performed using regional anesthesia, without preoperative sedatives, to facilitate the mother's conscious birth experience, reduce the need for neonatal resuscitation, and promote skin-to-skin contact immediately after birth between the mother and newborn. The VR can be designed to be an interacting and emotionally engaging environment that can stimulate emotionally related hormones. In stressful situations as CS, VR can generate a relaxation state that improves the surgery outcomes.

DETAILED DESCRIPTION:
The application of VR varies widely according to the purpose of its use. It is widely used for medical education, pain relief, posttraumatic stress, gait rehabilitation in Parkinson's disease patients, anxiety, and stress.

ELIGIBILITY:
Inclusion Criteria:

* female from 25 to 35 years
* post cesarean section

Exclusion Criteria:

* neurological problems
* musculoskeletal disorders

Ages: 25 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — problem is cesarean section which is happening in females only
Enrollment: 80 (Actual)
Dates: Start 2024-10-20 (Actual); Primary Completion 2025-04-02 (Actual); Study Completion 2025-07-20 (Actual)

PRIMARY OUTCOMES:
hand held dynamometer | 2 month
  isokinetic dynamometer
  hand held dynamometer hand held dynamometer used to measure the abdominal muscle strength, endurance and fatidue

SECONDARY OUTCOMES:
rectus diastasis test | 2 month
  manual test used to determine the separation between two recti

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo university, Cairo, Egypt